CLINICAL TRIAL: NCT05823532
Title: Targeting Inflammation-Induced Changes in Brain Reward Signaling and Motivational Deficits in Patients With Schizophrenia Using an Anti-Inflammatory Challenge.
Brief Title: Anti-Inflammatory Challenge in Schizophrenia
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, David Goldsmith, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: STUDY00004430; R01MH131910-01 (NIH)
Record Dates: First submitted 2023-02-08; First posted 2023-04-21 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Schizophrenia
Keywords: Inflammation; Reward-related Brain Regions
MeSH Terms: conditions — Schizophrenia; Inflammation | interventions — Infliximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Infliximab (Experimental): Subjects will be stratified by sex and randomized prior to this visit in preparation for the infusion. Vitals and safety labs will be drawn at this visit as well as urine testing for drugs of abuse and pregnancy testing for all biological females. Patients will receive breakfast followed by a double-blinded infusion of infliximab (5mg/kg body weight) in the GCSTA Clinical Research Center at Emory University Hospital. The infusion will last 3 hours, and subjects will be monitored during the infusion and for one hour after completion for the possible development of anaphylaxis, which occurs in less than 1% of patients receiving an initial dose of infliximab
  Interventions: Drug: Infliximab
- Placebo (Placebo Comparator): Subjects will be stratified by sex and randomized prior to this visit in preparation for the infusion. Vitals and safety labs will be drawn at this visit as well as urine testing for drugs of abuse and pregnancy testing for all biological females. Patients will receive breakfast followed by a double-blinded infusion of saline in the GCSTA Clinical Research Center at Emory University Hospital. The infusion will last 3 hours, and subjects will be monitored during the infusion and for one hour after completion for the possible development of anaphylaxis, which occurs in less than 1% of patients receiving an initial dose of infliximab
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Infliximab — Infliximab has FDA approval for the treatment of rheumatoid arthritis and inflammatory bowel syndrome. The current proposal represents the use of infliximab as an experimental tool to dissect the role of inflammatory processes leading to changes in brain reward circuitry and changes in specific symptom domains.
  Double-blinded infusions of infliximab will be administered in the GCTSA Clinical Research Center, located at Emory University Hospital. Independent pharmacists will dispense either infliximab or placebo in a 250ml saline bag according to a computer-generated randomization list provided by the study pharmacist.
  Arms: Infliximab
Drug: Placebo — Double-blinded infusions of saline will be administered in the GCTSA Clinical Research Center, located at Emory University Hospital. Independent pharmacists will dispense either infliximab or placebo in a 250ml saline bag according to a computer-generated randomization list provided by the study pharmacist.
  Arms: Placebo

SUMMARY:
This research project will explore negative symptoms of schizophrenia, such as motivational deficits, by examining the relationship between inflammation and reward-related brain regions. To accomplish this, we will administer a single infusion of either the anti-inflammatory medication infliximab or placebo (n=10 per group) to patients with high inflammation.

This study is important because schizophrenia can be a chronic and debilitating neuropsychiatric disorder and negative symptoms are some of the most difficult aspects of schizophrenia associated with worst functional outcomes. These symptoms do not typically respond to antipsychotic therapies, and as such, there are no current medications to treat negative symptoms.

DETAILED DESCRIPTION:
This research project will explore negative symptoms of schizophrenia, such as motivational deficits, by examining the relationship between inflammation and reward-related brain regions. To accomplish this, we will administer a single infusion of either the anti-inflammatory medication infliximab or placebo (n=10 per group) to patients with high inflammation.

This study is important because schizophrenia can be a chronic and debilitating neuropsychiatric disorder and negative symptoms are some of the most difficult aspects of schizophrenia associated with worst functional outcomes. These symptoms do not typically respond to antipsychotic therapies, and as such, there are no current medications to treat negative symptoms.

Study procedures include 9 separate visits as follows:

1. Pre-screening Visit which includes questions about mood and negative symptoms of schizophrenia, blood sampling to measure CRP which is a marker of inflammation, a urine drug screen (UDS) and urine testing for pregnancy in all biological women (approx. 1-2 hours).
2. Screening Visit which includes assessing for adverse events, more detailed questions about symptoms, a physical exam, blood draw for medical safety screening labs, magnetic resonance imaging (MRI) safety screening questionnaire, instruction and practice playing a computer game where the participant can earn money, and an electrocardiogram (EKG) to make sure the patient's heart is healthy.
3. Baseline Visit which includes assessing for adverse events, behavioral assessments, blood sampling for medical safety screening labs and research labs, functional magnetic resonance imaging (fMRI) scan where participant plays a computer game where s/he can earn extra money. Randomization to the study drug, Infliximab, or a placebo (approx. 5-6 hours).
4. Infusion Visit which includes assessing for adverse events, blood draw for safety screening labs, UDS and pregnancy testing, and infusion of the study drug, Infliximab, or a placebo (approx. 5 hours).
5. 24-hr Post Infusion Visit which includes behavioral assessments, vital signs, safety labs, and assessing for adverse events (approx. 1-2 hours).
6. 3-day Post Infusion Visit which includes assessing for adverse events, behavioral assessments, vital signs, safety labs (approx. 1-2 hours)
7. 7-day Post Infusion Visit which includes assessing for adverse events, behavioral assessments, vital signs and safety labs (approx. 1-2 hours)
8. 14-day Post Infusion Visit which includes assessing for adverse events, blood draw for safety labs, urine pregnancy and drug testing, fMRI scan and a lumbar puncture for cerebrospinal fluid (CSF)(approx. 6-7 hours)
9. One-month Follow-up Safety Check-in which includes a phone call to assess for adverse (approx. 10-15 minutes).

Approximately 60 subjects will be consented and prescreened in order to obtain complete data on 20 medically stable, male, and female adult subjects with schizophrenia or schizoaffective disorder at the Grady Behavioral Health Clinic.

Blood will be collected across multiple visits, some of which will be stored for future research use.

Written informed consent will be obtained in a private office at the Grady Behavioral Health Clinic. All aspects of the study will be reviewed and a discussion will occur to make sure the participant is aware of all study details. Should a subject agree to study participation, s/he will be given a copy of the informed consent for their records. In addition, the process of informed consent will continue throughout the course of each study visit to be sure the participant is fully aware of all procedures. If the participant has a legally authorized representative (LAR), the LAR will be required to attend the initial prescreening visit and sign the informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Men or women, 18-45 years of age with a primary diagnosis of Diagnostic and Statistical Manual of Mental Disorders (DSM-V) schizophrenia or schizoaffective disorder;
* Willing and able to give written informed consent;
* Plasma CRP 3mg/L;
* Significant motivational deficit as reflected by a score >17 on the Motivation and Pleasure Domain of the Brief Negative Symptom Scale. Of note, for patients who exhibit CRP>10mg/L, additional CRP testing will be conducted at 2-week intervals as per American Heart Association/ Center for Disease and Control Prevention guidelines to establish stability and rule out acute inflammation/infection (along with physical exam and laboratory testing).
* Patients must also have a negative urine drug screen at all study visits.

Exclusion Criteria:

* Any autoimmune disorder (as confirmed by laboratory testing);
* History of tuberculosis infection as determined by QuantiFERON Gold or high risk of tuberculosis exposure;
* Active hepatitis B or C infection or human immunodeficiency virus infection (as established by laboratory testing);
* History of any type of cancer;
* History of fungal infection;
* History of recurrent viral or bacterial infections;
* Unstable cardiovascular (including evidence of congestive heart failure as determined by physical examination and laboratory testing), endocrinologic, hematologic, hepatic, renal, and neurological disease (as determined by physical examination and laboratory testing);
* Demyelinating brain disease and/or a concerning structural abnormality seen on MRI;
* Substance abuse/dependence within 6 months of study entry (as determined by MINI and urine drug screen);
* Primary diagnosis of mood or anxiety disorder (i.e., major depressive disorder, bipolar disorder, post-traumatic stress disorder) as determined by the International Neuropsychiatric Interview for Schizophrenia and Psychotic Disorders (MINI).
* Active suicidal ideation or plan;
* An active eating disorder;
* A history of cognitive disorder or Mini-Mental State Exam (MMSE) < 24 (indicating cognitive impairment);
* Pregnancy or lactation;
* Treatment with clozapine (given increased risk of neutropenia/agranulocytosis);
* Women of childbearing potential who are not using a medically accepted means of contraception;
* Known allergy to murine products or other biologic therapies;
* Previous organ transplant;
* Administration of any modified live virus vaccine within one month of study entry, during the study, and for at least one month after the final study visit;
* Oral glucocorticoids, immunosuppressive drugs (e.g. anti-cytokine therapies or methotrexate), or any other drugs targeting the immune system within 6 months of baseline;
* Chronic use of non-steroidal anti-inflammatory agents (NSAIDs; excluding 81mg of aspirin), glucocorticoid-containing medications, or minocycline or non-prescription supplements with known or suspected anti-inflammatory properties (e.g. fish oil supplements, curcumin, pre- or probiotics) within 2 weeks of baseline or at any time during the study;
* Use of non-steroidal anti-inflammatory agents (NSAIDs), and glucocorticoid medications at any time during the study;
* Any contraindication to MRI. Due to the high co-morbidity between schizophrenia and mood/anxiety disorders, the study team plans to include patients with these diagnoses as long as schizophrenia is the primary diagnosis.
* Subjects may be taking psychotropic medications at the time of the study (including antipsychotics, antidepressants, mood stabilizers, and benzodiazepines) but may have no psychotropic medication changes for one month before study enrollment or during participation in the study. Patients with stable medical conditions and on medications for those conditions will not be excluded. No patient will be removed from antipsychotic treatment for this study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-04-18 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Changes in Monetary Incentive Delay Task (MID) | Study visits: 1-3 days before intervention and 6 weeks post-intervention
  Change in Bold Oxygen Level Dependent (BOLD) Activation in the Ventral Striatum during "Win" Monetary Incentive Delay (MID) Task between Infliximab and Placebo (time frame: 1-3 days between first scan and intervention and then 2 weeks between intervention and repeat scan). Activation response in ventral striatum in response to reward anticipation: Infliximab (vs placebo)-treated patients will exhibit a) increased activation in ventral striatum in response to reward. Mixed-effects models for repeated measures (MMRM) will first be employed to examine effects of group (infliximab vs. placebo), time and their interaction on blood oxygenation level-dependent (BOLD) signals (an index of regional brain activation) using a Region-of-Interest (ROI) approach.
Changes in Effort Based Decision Making Task (EBDM) | Study Visits :1-3 days before intervention,3 days post intervention, 1 week and 2 weeks post-intervention
  Changes in BOLD Activation response in anterior insula in response to increasing effort between Infliximab and Placebo (time frame: 1-3 days between first scan and intervention and then 2 weeks between intervention and repeat scan). Activation response in insula in response to increasing effort: Infliximab (vs placebo)-treated patients will exhibit a) decreased activation in anterior insula in response to effort.
  Mixed-effects models for repeated measures (MMRM) will first be employed to examine effects of group (infliximab vs. placebo), time and their interaction on BOLD signals (an index of regional brain activation) using a Region-of-Interest (ROI) approach.
Changes in C-Reactive Protein (CRP) | Study Visits :1-3 days before intervention, immediately after the intervention, 1 day post-intervention, 3 days, 1 week and 2 weeks post-intervention
  30ml study bloods per visit will be collected by venipuncture into EDTA-containing vacutainer tubes using standard sterile technique. Plasma for the evaluation of plasma concentrations of CRP will be obtained by centrifugation of whole blood at 1000 x g for 10 minutes at 4 C.
  Plasma CRP will be assessed with a high sensitivity turbidimetric assay. Assay sensitivity is rated at 0.18 mg/L, range of measure is 0.2 to 80 mg/L and functional sensitivity (at 20% CV) is 0.2 mg/L.
Changes in Brief Negative Symptom Scale (BNSS) | Study Visits :1-3 days before intervention,3 days post intervention, 1 week and 2 weeks post-intervention
  Infliximab (vs placebo) -treated patients will record their performance on the BNSS Motivation and Pleasure domain score.
  The BNSS is a 13-item scale designed for research studies in response to the 2005 National Institute of Mental Health (NIMH) consensus development conference on negative symptoms of schizophrenia.The BNSS measures the five commonly accepted domains of negative symptoms: blunted affect, alogia, asociality, anhedonia, and avolition. Items are scored on a 0 to 6 scale, with 0 indicating the symptom is absent and 6 indicating the symptom is severe. Items are summed for a total score that ranges between 0 and 78.

SECONDARY OUTCOMES:
Changes in Performance on the Effort Expenditure for Reward Task | Study Visits :1-3 days before intervention,3 days post intervention, 1 week and 2 weeks post-intervention
  Infliximab (vs placebo) -treated patients will be evaluated on their performance on the EEfRT.
  Assessment of reward motivation will be accomplished using an fMRI-adapted version of the EEfRT task. During each trial, subjects are presented with a choice between two levels of task difficulty, a High Effort option and a Low Effort option, which require different amounts of speeded manual button pressing for differing levels of monetary reward. The reward magnitude for a No Effort option remains constant , while the reward magnitude for the High Effort option will vary between 20%, 50%, 80%, and 100% of the subjects max effort (set for each individual prior to scan). The task will use a rapid event-related design with an exponential jitter between trials drawn in order to optimize hemodynamic response function estimation. Responses will be made using MRI-compatible button-boxes and images will be presented on a rear projection screen visible with a mirror mounted on the head coil.
Changes in Positive and Negative Syndrome Scale (PANSS) | Study Visits :1-3 days before intervention,3 days post intervention, 1 week and 2 weeks post-intervention
  Infliximab (vs placebo) -treated patients will record their performance on the Positive and Negative Syndrome Scale (PANSS) The PANSS is the most commonly used measure of assessing the symptoms of schizophrenia. Seven items measure positive symptoms, seven measure negative symptoms, and sixteen measure general psychopathology symptoms. PANSS items are rated on a 7-point scale (1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, and 7=extreme); because the absence of symptoms is equal to 1 point, the lowest possible total score on both PANSS scales is 7.
Changes in Motivation and Pleasure Scale (MAPS-SR) | Study Visits :1-3 days before intervention,3 days post intervention, 1 week and 2 weeks post-intervention
  The MAPS-SR is a 15-item self-report scale that has demonstrated good convergent validity with the clinician-rated Motivation and Pleasure scale of the Clinical Assessment Interview for Negative Symptoms (CAINS). The scale has four subscales that include ratings of social pleasure, recreational or work pleasure, feelings and motivations about close, caring relationships, and motivation and effort to engage in activities, corresponding to the CAINS subscales of deficits in motivation and pleasure and deficits of expression.
  (MAP-SR) Six items tap consummatory and anticipatory pleasure related to social and recreational or work domains. Six items tap feelings and motivations to be around family, romantic partners, and friends. The remaining six items tap motivation and effort to engage in activities. All items are rated on a 5-point Likert scale; higher scores reflect greater pathology after reverse scoring for items 8, 10, and 12.
Changes in Calgary Depression Scale for Schizophrenia (CDSS) | Study Visits :1-3 days before intervention, immediately after the intervention, 1-day post-intervention, 3 days, 1 week and 2 weeks post-intervention
  The CDSS is a clinician-administered, 9-item rating scale designed for the assessment of depressive symptoms in schizophrenia. Depressive symptoms are highly prevalent in patients with schizophrenia and may lead to a higher burden of disease. It is reliable, valid, and able to distinguish depressive symptoms from negative symptoms and extrapyramidal symptoms.
Changes in Inflammatory markers changes: IL-1 | Study Visits :1-3 days before intervention, immediately after the intervention, 1-day post-intervention, 3 days, 1 week and 2 weeks post-intervention
  Customized Fluorokine MAP Multiplex Human Biomarker Panels (R&D Systems, Minneapolis, MN) will be used to measure plasma Interleukin (IL)-1 receptor antagonist. This inflammatory marker was chosen based on its reliable changes in psychiatric illness and/or their relationship to symptoms of anhedonia and corticostriatal function.
Changes in Inflammatory markers changes: IL-6 | Study Visits :1-3 days before intervention, immediately after the intervention, 1-day post-intervention, 3 days, 1 week and 2 weeks post-intervention
  Customized Fluorokine MAP Multiplex Human Biomarker Panels (R&D Systems, Minneapolis, MN) will be used to measure plasma IL-10. This inflammatory marker was chosen based on its reliable changes in psychiatric illness and/or their relationship to symptoms of anhedonia and corticostriatal function.
Changes in Inflammatory markers changes: IL-10 | Study Visits :1-3 days before intervention, immediately after the intervention, 1-day post-intervention, 3 days, 1 week and 2 weeks post-intervention
  Customized Fluorokine MAP Multiplex Human Biomarker Panels (R&D Systems, Minneapolis, MN) will be used to measure plasma IL-10. This inflammatory marker was chosen based on its reliable changes in psychiatric illness and/or their relationship to symptoms of anhedonia and corticostriatal function.
Changes in Inflammatory markers changes: Soluble IL-6R | Study Visits :1-3 days before intervention, immediately after the intervention, 1-day post-intervention, 3 days, 1 week and 2 weeks post-intervention
  Customized Fluorokine MAP Multiplex Human Biomarker Panels (R&D Systems, Minneapolis, MN) will be used to measure plasma soluble IL-6R. This inflammatory marker was chosen based on its reliable changes in psychiatric illness and/or their relationship to symptoms of anhedonia and corticostriatal function.
Changes in Inflammatory markers changes: Tumor necrosis factor (TNF) | Study Visits :1-3 days before intervention, immediately after the intervention, 1 day post-intervention, 3 days, 1 week and 2 weeks post-intervention
  Customized Fluorokine MAP Multiplex Human Biomarker Panels (R&D Systems, Minneapolis, MN) will be used to measure plasma TNF This inflammatory marker was chosen based on its reliable changes in psychiatric illness and/or their relationship to symptoms of anhedonia and corticostriatal function.
Changes in Inflammatory markers changes: sTNFR2 | Study Visits :1-3 days before intervention, immediately after the intervention, 1-day post-intervention, 3 days, 1 week and 2 weeks post-intervention
  Customized Fluorokine MAP Multiplex Human Biomarker Panels (R&D Systems, Minneapolis, MN) will be used to measure plasma sTNFR2. This inflammatory marker was chosen based on its reliable changes in psychiatric illness and/or their relationship to symptoms of anhedonia and corticostriatal function.
Changes in Inflammatory markers changes: monocyte chemoattractant protein (MCP)-1 | Study Visits :1-3 days before intervention, immediately after the intervention, 1-day post-intervention, 3 days, 1 week and 2 weeks post-intervention
  Customized Fluorokine MAP Multiplex Human Biomarker Panels (R&D Systems, Minneapolis, MN) will be used to measure plasma monocyte chemoattractant protein (MCP)-1. This inflammatory marker was chosen based on its reliable changes in psychiatric illness and/or their relationship to symptoms of anhedonia and corticostriatal function.
Changes in Quality-of-Life Enjoyment and Satisfaction Questionnaire Short Form | Study Visits :1-3 days before intervention, 1 week and 2 weeks post-intervention
  The Q-LES-Q-SF evaluates general activities that are assessed in the longer form of the Q- LES-Q. Each item uses a 5-point scale ranging from 1 (very poor) to 5 (very good). A total score is derived from 14 items with a maximum score of 70 and with higher scores indicating greater life satisfaction and enjoyment. Participants rate their satisfaction with the following domains of activity: physical health, feelings, work, household duties, school/course work, leisure time activities, and social relations.
Changes in The Calgary Depression Scale for Schizophrenia (CDSS) | Study Visits :1-3 days before intervention, 1 week and 2 weeks post-intervention
  The Calgary Depression Scale for Schizophrenia (CDSS) is a nine-item structured interview scale that was designed in 1990 specifically to assess depression independently of symptoms of psychosis in schizophrenia.
  Point scores of all nine items are summed to obtain the CDS depression score. A score higher than 6 has an 82% specificity and 85% sensitivity for predicting the presence of a major depressive episode.
Changes in WHO Disability Assessment Schedule (WHODAS) | Study Visits :1-3 days before intervention, 1 week and 2 weeks post-intervention
  The World Health Organization Disability Assessment Schedule (WHODAS 2.0) is a practical, generic assessment instrument that can measure health and disability at population level or in clinical practice (World Health Organization (WHO).
  The first score is determined using "item-response-theory" (IRT), where it considers multiple levels of difficulty for each WHODAS 2.0 item (1-36). This type of scoring for WHODAS 2.0 allows for more fine-grained analyses that make use of the full information of the response categories for comparative analysis across populations or subpopulations. It takes the coding for each item response as "none", "mild", "moderate", "severe" and "extreme" separately, and then summarizes the score by differentially weighting the items and the levels of severity. Converting the summary score into a metric ranging from 0 to 100 (where 0 = no disability; 100 = full disability)

CONTACTS AND LOCATIONS:
Overall Officials: David R Goldsmith, MD, Principal Investigator — Assistant Professor
Locations (2):
- United States (2):
  - Grady Memorial Hospital, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
Phenotypic, biomarker, and neuroimaging data may be shared by request to the PI two years after publication of the primary study results.
Supporting Information: Study Protocol, SAP
Time Frame: Two years after publication of the primary study results with no specified end date
Access Criteria: Access criteria decisions will be made by the PI, via communication with him.